CLINICAL TRIAL: NCT00258947
Title: Take Evaluation and Safety of Smallpox Vaccine (LISTER Strain) in Naïve Healthy Adults.
Brief Title: Evaluation of Take and Safety of a Smallpox Vaccine in Healthy Young Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VVL04
Record Dates: First submitted 2005-11-24; First posted 2005-11-28 (Estimated); Last update posted 2012-02-01 (Estimated); Status verified 2012-01

CONDITIONS: Smallpox; Poxvirus Infection
Keywords: Smallpox; Orthopoxvirus; Poxvirus; Vaccina Virus; LISTER Strain; Bioterrorism
MeSH Terms: conditions — Smallpox; Poxviridae Infections | interventions — Smallpox Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: Smallpox vaccine, LISTER strain, from chick embryo cells

SUMMARY:
Primary Objective:

To estimate the smallpox vaccination take rate in healthy young adults not previously vaccinated with a smallpox vaccine.

Secondary Objectives:

To describe antibody response to vaccination and evaluate the take for each subject at various timepoints for each batch and pooled batches and to evaluate local signs, symptoms, and overall safety in healthy young adults not previously vaccinated with a smallpox vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 25 years on the day of screening
* Informed consent form signed
* Able to attend all scheduled visits and to comply with all trial procedures
* For a woman, inability to bear a child or negative serum pregnancy test performed at screening (Visit 01)
* Subject entitled to national social security
* Subject registered in the French file of healthy volunteers in clinical trials
* For a woman of child-bearing potential: use of an effective method of contraception (hormonal or barrier method) from at least 3 months prior to screening to 3 months following trial vaccination
* For a woman, inability to bear a child or negative urine pregnancy test.

Exclusion Criteria:

* Previous smallpox vaccination confirmed by vaccination record or typical scar
* Participation in another trial in the 3 months before or during the trial period
* Acute intercurrent or chronic illness during the trial
* Breast-feeding
* Allergy or sensitivity to any known components of vaccinia immune globulin or previous reaction to immunoglobulins or trial vaccine
* Congenital or acquired immunodeficiency or immunosuppressive therapy or any treatment including corticosteroids
* Treatment with antiviral drugs within 1 month before vaccination
* History of organ or bone marrow transplant or skin disorders
* Personal or family history of autoimmune disease or cardiac disease, including cardiac risk factors
* History or current central nervous system disease
* Ongoing acute infectious disease
* Blood or blood-derived products received in the past 6 months
* Any vaccination with a live-attenuated vaccine within the 60 days or other vaccines within 40 days preceding the trial vaccination
* Vaccination planned in the 8 weeks following the trial vaccination
* Planned or foreseeable close contact after vaccination with infants less than 12 months, or with immuno-suppressed persons, pregnant and/or lactating woman, or practice of contact or water sports after vaccination before the crust separates
* Skin wound near the vaccination site
* Apparent lack of personal hygiene
* Subject deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized without his/her consent
* HIV, hepatitis B or hepatitis C seropositivity (screening tests)
* Abnormal lab values for hematological parameters or cardiac enzyme (screening tests)
* Feverish illness (oral temperature >=37.5°C, rectal equivalent temperature >=38.0°C) on the day of vaccination.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 230 (Actual)
Dates: Start 2005-09; Primary Completion 2006-12 (Actual); Study Completion 2007-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc
Locations (6):
- France (6):
  - Gières
  - Lagord
  - Montpellier
  - Paris
  - Poitiers
  - Rouen

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com